CLINICAL TRIAL: NCT02522156
Title: Looming Vulnerability and Smoking Cessation Attempts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University (Other)
Responsible Party: Principal Investigator, David A. F. Haaga, Professor of Psychology, American University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: American_University
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Looming Vulnerability Induction (Experimental): Four audiotape-guided imagery exercises, each lasting about 3 minutes:
  * Conveyor Belt: Places the participants in a dimly-lit factory, in which they are being carried along faster and faster on a conveyor belt as they smoke. This conveyor belt is described as ultimately leading to the diagnosis of lung cancer.
  * Office Building: Places participants in an office all alone, watching calendar pages fly off the wall. As participants smoke and time progresses, participants are meant to feel their lungs withering away and their heart beat becoming weaker and weaker.
  * Train Tracks: Set in the open plains on top of a set of railroad tracks. As participants smoke, a train heading directly towards them gains speed.
  * Clock Ticking: In this timing exercise, participants are instructed to imagine terrible health consequences related to smoking coming closer and closer to them as they smoke. Participants are asked to keep track of time for a period of three minutes.
  Interventions: Behavioral: Looming Vulnerability Induction
- Control (Placebo Comparator): Four audiotape-guided imagery exercises, as follows:
  * Escalator (parallel to "conveyor belt" above): Takes place in an empty mall in the morning. The participants imagine they are slowly and steadily being carried by the escalator until they reach the top.
  * Metro (parallel to "office building"): Involves riding public transportation while reading a magazine, steadily flipping the pages.
  * Driving (parallel to "Train Tracks"): Involves driving a car. The car in this case moves steadily with no traffic hindrances that would cause a reduction of speed.
  * Human Clock (parallel to "Clock Ticking"): Another timing exercise. In this case, the participants receive instruction to pretend they are a human clock.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Looming Vulnerability Induction — guided imagery aimed at inducing smoking cessation attempts. See description of the looming vulnerability arm.
  Arms: Looming Vulnerability Induction
Behavioral: Control — Neutral guided imagery scenarios making no reference to smoking.
  Arms: Control

SUMMARY:
Almost one-fifth of US adults are current cigarette smokers. To make further progress in lowering prevalence, it would help to increase the proportion of smokers attempting to quit. This application tests a novel approach to motivating smokers to quit, based on an empirically supported theory of anxiety. The approach uses guided imagery to increase smokers' sense of urgency about preventing the negative health consequences of smoking.

DETAILED DESCRIPTION:
Approach Participants and Eligibility Criteria

The investigators plan to enroll 290 participants, recruited via newspaper, radio, and online ads, flyers distributed in the community, and letters to healthcare providers. Ads will recruit adults who smoke at least 10 cigarettes/day and are willing to participate in two sessions four weeks apart but will not mention smoking cessation.

Prospective participants must meet the following criteria at a phone screen:

1. Adults (age 18 or older).
2. Daily cigarette smokers (at least 10 cigarettes per day).
3. Total score of 5 or below on the Modified Mini Screen and score of 0 on the suicidality item.
4. Fluent in English.
5. Not planning to leave the Washington, DC area in the next month.

The Modified Mini Screen (MMS) is a safety precaution for the looming vulnerability induction, which on average increases state anxiety. Those scoring 6 or higher on the MMS are considered at moderate to high risk of having anxiety, mood, or psychotic disorders. The MMS is a modification of the MINI and appears to work equally well for men and women and for Caucasians and African Americans; the investigators are using the lowest (most conservative) cutoff score recommended on the basis of research validating the MMS against a full diagnostic interview (SCID). Prospective participants excluded on this basis will be offered therapy in a departmental training clinic, as well as alternate local referrals, outside the context of this research project.

Fluency in English is necessary for valid completion of our assessments. Planning to remain in the metropolitan area should help to lower the attrition rate.

Procedure

Eligible participants who choose to enroll in the study will be scheduled for an in-person assessment and imagery experiment. The following chart shows measures completed at each assessment:

Measure Experiment 4-week follow-up Expired air CO X X State anxiety (VAS) X (pre/post imagery induction) Demographics X Smoking and smoking cessation history X Nicotine Dependence (FTND) X X Visualization ability (VVIQ) X Contemplation Ladder X X Stage of change algorithm X X Current (past month) smoking rate X X Self-efficacy (SSEQ) X X Outcome expectancies (SCQ-A) X X Most accessible outcome expectancy (SGO) X X Vividness rating of imagery X Perception of health consequences of smoking as looming (CSCLS-P) X Quit attempt (>= 24 hours) X Description of quit attempt methods used, length, etc. X Sensation Seeking (SSS-V) X

First session: Baseline assessment and experiment on looming vulnerability induction. After completing informed consent, participants will complete an expired air CO test to corroborate smoker status (>= 9 ppm). If smoker status is not confirmed, they will be paid for their time and excused as ineligible. Participants who are eligible and interested will complete baseline measures in one of four random orders:

Visual Analogue Scale (VAS) for state anxiety. State anxiety will be measured with a single-item VAS in which the participant makes a mark along a 100 mm horizontal line anchored by the phrase "Not at All" at the left (0) and "Extremely" at the right end (100), with the word "Anxious" printed above the line in the middle; the score is the number of millimeters from the left end at which the participant made the mark. VAS measures have proven useful as indicators of state anxiety in smoking research.

Demographics, smoking history, quitting history, and current (past month) smoking rate will be measured with brief, face-valid questionnaires. The investigators have used in previous studies a 10-item measure of current smoking rate, years of smoking, and length of longest and most recent attempts to quit smoking. This measure is similar to, but a bit more detailed than, the Active Smoking Questionnaire downloadable from the NCI website. It will be adapted for this study to assess e-cigarette use, which is rapidly increasing, with at least one-third of US adult smokers having ever used e-cigarettes.

Nicotine dependence will be indexed by the Fagerstrom Test of Nicotine Dependence (FTND17), a 6-item scale with moderate internal consistency and predictive validity in relation to abstinence in studies of varenicline.

Visualization ability will be measured with the revised Vividness of Visual Imagery Questionnaire (VVIQ2). Respondents are asked to form images of specific scenes and rate their vividness. Validity data are favorable. For example, high scorers are more likely to notice changes made to pictures they are shown.

Sensation seeking will be measured with the revised Sensation Seeking Scale-V. This forced-choice self-report measure shows high internal consistency and extensive evidence of concurrent validity in relating to attitudinal and behavioral criteria theoretically associated with sensation seeking.

Contemplation of quitting will be measured in two ways. The Contemplation Ladder (CL) consists of a ladder with rungs labeled 1 to 10. The lowest score (0, below the bottom rung) represents "no thought of quitting", whereas the highest score (10) reflects "taking action to quit (e.g., cutting down, enrolling in a program)". In a national population-based study of smokers not initially interested in quitting immediately, CL scores predicted making a quit attempt in response to an intervention. Also, self-reports will be used to stage smokers according to an algorithm (no intention to quit within next six months = precontemplators; intending to quit in next six months but not next 30 days = contemplators; intending to quit in next 30 days = preparers).

Self-efficacy will be measured with the Smoking Self-Efficacy Questionnaire (SSEQ), a 17-item self-report measure of confidence in one's ability to resist temptation to smoke in various high-risk situations. SSEQ scores have been shown to predict length of time to first relapse after a smoking cessation attempt.

Outcome expectancies for smoking will be measured in two ways. First, on the premise that highly accessible expectancies regarding smoking may be the most influential in determining smoking-related behavior, the "Self-Generated Outcome (SGO)" test calls for completion of the stem "When I smoke cigarettes, I expect to …..", and coding is based solely on the first response. Scores are sensitive to current mood and to smoking status. Second, the Smoking Consequences Questionnaire-Adult (SCQ-A) is a well-validated 55-item self-report measure of expected consequences of cigarette smoking.

Experimental manipulation of looming vulnerability. After completing baseline measures, participants will be randomly assigned to either the looming condition or the control condition (using a pre-selected random order generated via www.randomizer.org, with the condition unknown to the experimenter until this point).

The randomization will be stratified by sex and by whether the participant had ever made an attempt to quit smoking previously.

The imagery scenarios in each of the conditions (looming or control) will be the ones used in McDonald et al. presented in one of four random orders.

Posttest measures: manipulation check and hypothesized mediator: After the imagery exercises, participants will complete a second state anxiety VAS as an immediate manipulation check, along with a rating of the vividness of the imagery. They will then complete the CSCLS-P (see description and validity evidence in preliminary studies section above) to measure their perception of the physical health consequences of smoking as looming threats. This measure will be tested as a hypothesized mediator of the effects of the imagery induction on quit attempts.

Advice to quit. At the completion of the assessments, the experimenter will give the participant (regardless of experimental condition) a handout containing brief advice to quit smoking, along with written information about (a) quitnet.com as a free site they could use to obtain community support and extensive information concerning nicotine replacement therapy, medications, behavioral methods for coping with high-risk situations, preparation for quit date, and more, as well as (b) the telephone-based counseling provided for free via 1-800-QUIT-NOW.

Four-week follow-up assessment. Four weeks later there will be a second session, at which participants will complete the CL and algorithm measures as indicators of contemplation status as well as expectancy measures. Participants will also report on smoking rates and quit attempts since the first experimental session. Quit attempts are the primary outcome, but the investigators also consider changes in smoking rate meaningful. If participants claim to have made a quit attempt, they will be asked for the duration of the attempt and whether it is still in effect (i.e., whether they are currently abstinent, including no e-cigarette use given that the health implications of switching to e-cigarette use remain uncertain. Participants will complete an expired air CO test, and abstinence will be considered corroborated by a reading of < 8 ppm.

To minimize demand effects, the four-week follow-up session will always be conducted by a research assistant who (a) did not conduct time 1 assessments and (b) is masked to the experimental condition of the participant.

The protocol at follow-up will be as follows:

1. Interview regarding any quit attempts of at least 24 hours since the lab experiment. If there have been one or more such attempts, details will be sought concerning how long the attempt lasted, whether it is ongoing, and what methods were used. The remaining measures will be retests from baseline:
2. Current smoking rate.
3. Nicotine dependence.
4. Expired air CO reading.
5. Contemplation of quitting smoking.
6. Self-efficacy
7. Outcome expectancies.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age 18 or older).
2. Daily cigarette smokers (at least 10 cigarettes per day).
3. Fluent in English. -

Exclusion Criteria:

1. planning to leave the Washington, DC area in the next month.
2. Total score > 5 on the Modified Mini Screen measure of risk for anxiety or mood disorders
3. Score > 0 on the suicidality item (#4) of Modified Mini Screen -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2016-02; Primary Completion 2019-07 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Quit attempt | 4-week follow-up
  yes/no, whether or not the participant made a 24-hour (or longer) quit attempt between the date of the main experiment and the date of the 4-week follow-up assessment.

SECONDARY OUTCOMES:
Abstinence | 4-week follow-up
  CO-corroborated abstinence from smoking at 4-week follow-up.
Smoking rate | 4-week follow-up
  past-month average daily smoking rate
Contemplation of quitting | 4-week follow-up
  Contemplation ladder score
self-efficacy (Smoking Self-Efficacy Questionnaire; SSEQ) | 4-week follow-up
  confidence in ability to quit smoking
outcome expectancies (Smoking Consequences Questionnaire-Adult; SCQ-A) | 4-week follow-up
  expected consequences of cigarette smoking

CONTACTS AND LOCATIONS:
Locations (1):
- American University, Washington D.C., District of Columbia, United States